CLINICAL TRIAL: NCT02184195
Title: A Phase III, Randomised, Double Blind, Placebo Controlled, Multicentre Study of Maintenance Olaparib Monotherapy in Patients With gBRCA Mutated Metastatic Pancreatic Cancer Whose Disease Has Not Progressed on First Line Platinum Based Chemotherapy
Brief Title: Olaparib in gBRCA Mutated Pancreatic Cancer Whose Disease Has Not Progressed on First Line Platinum-Based Chemotherapy
Acronym: POLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D081FC00001; 2014-001589-85 (EudraCT Number)
Record Dates: First submitted 2014-06-06; First posted 2014-07-09 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-06

CONDITIONS: Germline BRCA1/2 Mutations and; Metastatic Adenocarcinoma of the Pancreas
Keywords: BRCA, metastatic adenocarcinoma pancreas, maintenance olaparib monotherapy, first line platinum chemotherapy, pancreatic cancer, PARP inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib (Experimental): Olaparib tablets po. 300 mg twice daily
  Interventions: Drug: Olaparib
- Placebo (Placebo Comparator): Placebo tablets twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olaparib — Tablet -100mg
  Arms: Olaparib
Drug: Olaparib — Tablet-150mg
  Arms: Olaparib
Drug: Placebo — Match Olaparib 100mg placebo
  Arms: Placebo
Drug: Placebo — Match Olaparib 150mg placebo
  Arms: Placebo

SUMMARY:
A Phase III, Randomised, Double Blind, Placebo Controlled, Multicentre Study of Maintenance Olaparib Monotherapy in Patients with gBRCA Mutated Metastatic Pancreatic Cancer whose Disease Has Not Progressed on First Line Platinum Based Chemotherapy

DETAILED DESCRIPTION:
Approximately 145 patients will be randomised using an Interactive Voice Response System /Interactive Web Response System (IVR/IWR system) in a 3:2 ratio (Olaparib:placebo) to the treatments as specified below:

* Olaparib tablets p.o. 300 mg twice daily
* Matching placebo tablets p.o. twice daily Eligible patients will be those patients with pancreas cancer previously treated for metastatic disease who have not progressed following completion of at least 16 weeks (can be more) of first line platinum-based chemotherapy. All patients must have a known deleterious or suspected deleterious germline BRCA mutation to be randomised; this may have been determined prior to enrolment into the study or may be assessed as part of the enrolment procedure for the study (via centrally provided MyriadIntegrated BRAC.

Patients will be randomised within 6 weeks after their last dose of chemotherapy (last dose is the day of the last infusion) and treatment started as soon as possible but no less than 4 and no more than 8 weeks of the last chemotherapy dose. At the time of starting protocol treatment, all previous chemotherapy treatment should be discontinued.

Following randomisation, patients will attend clinic visits weekly for the first 4 weeks of treatment (Days 8, 15, 22 and 29). Patients will then attend clinic visits every 4 weeks whilst on study treatment. Patients should continue to receive study treatment until objective radiological disease progression as per RECIST as assessed by the investigator and as long as in the investigator's opinion they are benefiting from treatment and they do not meet any other discontinuation criteria.

Once a patient has progressed the patient will be followed for second progression (PFS2) every 8 weeks and then survival until the final analysis.

ELIGIBILITY:
Key Inclusion Criteria

* Histologically or cytologically confirmed pancreas adenocarcinoma receiving initial chemotherapy for metastatic disease and without evidence of disease progression on treatment
* Patients with measurable disease and/or non-measurable or no evidence of disease assessed at baseline by CT (or MRI where CT is contraindicated) will be entered in this study.
* Documented mutation in gBRCA1 or gBRCA2 that is predicted to be deleterious or suspected deleterious
* Patients are on treatment with a first line platinum-based (cisplatin, carboplatin or oxaliplatin) regimen for metastatic pancreas cancer, have received a minimum of 16 weeks of continuous platinum treatment and have no evidence of progression based on investigator's opinion.
* Patients who have received platinum as potentially curative treatment for a prior cancer (eg ovarian cancer) or as adjuvant/neoadjuvant treatment for pancreas cancer are eligible provided at least 12 months have elapsed between the last dose of platinum-based treatment and initiation of the platinum-based chemotherapy for metastatic pancreas cancer.

Major Exclusion Criteria:

* gBRCA1 and/or gBRCA2 mutations that are considered to be non detrimental (eg, "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favour polymorphism" or "benign polymorphism" etc.)
* Progression of tumour between start of first line platinum based chemotherapy for metastatic pancreas cancer and randomisation.
* Cytotoxic chemotherapy or non-hormonal targeted therapy within 28 days of Cycle

  1 Day 1 is not permitted.
* Exposure to an investigational product within 30 days or 5 half lives (whichever is longer) prior to randomisation
* Any previous treatment with a PARP inhibitor, including Olaparib

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (17):
  - Research Site, Gilbert, Arizona
  - Research Site, Orange, California
  - Research Site, Stanford, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Commack, New York
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Australia (3):
  - Research Site, Campbelltown
  - Research Site, Randwick
  - Research Site, St Leonards
- Belgium (3):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Leuven
- Canada (4):
  - Research Site, London, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Toronto
- France (14):
  - Research Site, Amiens
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Clichy
  - Research Site, La Roche-sur-Yon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (11):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Dresden
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Schweinfurt
  - Research Site, Ulm
- Israel (9):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Zefir
- Italy (8):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Pescara
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
  - Research Site, Verona
- Research Site, Amsterdam, Netherlands
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (10):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Sabadell
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
  - Research Site, Zaragoza
- United Kingdom (8):
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Nottingham
  - Research Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- [Derived] Kindler HL, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, Bordia S, McGuinness D, Cui K, Locker GY, Golan T. Overall Survival Results From the POLO Trial: A Phase III Study of Active Maintenance Olaparib Versus Placebo for Germline BRCA-Mutated Metastatic Pancreatic Cancer. J Clin Oncol. 2022 Dec 1;40(34):3929-3939. doi: 10.1200/JCO.21.01604. Epub 2022 Jul 14. PMID 35834777
- [Derived] Amin S, Joo S, Nolte S, Yoo HK, Patel N, Byrnes HF, Costa-Cabral S, Johnson CD. Health-related quality of life scores of metastatic pancreatic cancer patients responsive to first line chemotherapy compared to newly derived EORTC QLQ-C30 reference values. BMC Cancer. 2022 May 20;22(1):563. doi: 10.1186/s12885-022-09661-7. PMID 35596182
- [Derived] Li N, Zheng H, Huang Y, Zheng B, Cai H, Liu M. Cost-Effectiveness Analysis of Olaparib Maintenance Treatment for Germline BRCA-Mutated Metastatic Pancreatic Cancer. Front Pharmacol. 2021 Apr 20;12:632818. doi: 10.3389/fphar.2021.632818. eCollection 2021. PMID 33959007
- [Derived] Zhan M, Zheng H, Yang Y, He Z, Xu T, Li Q. Cost-Effectiveness Analysis of Maintenance Olaparib in Patients with Metastatic Pancreatic Cancer and a Germline BRCA1/2 Mutation Based on the POLO Trial. Cancer Manag Res. 2020 Dec 16;12:12919-12926. doi: 10.2147/CMAR.S283169. eCollection 2020. PMID 33364840
- [Derived] Golan T, Kindler HL, Park JO, Reni M, Macarulla T, Hammel P, Van Cutsem E, Arnold D, Hochhauser D, McGuinness D, Locker GY, Goranova T, Schatz P, Liu YZ, Hall MJ. Geographic and Ethnic Heterogeneity of Germline BRCA1 or BRCA2 Mutation Prevalence Among Patients With Metastatic Pancreatic Cancer Screened for Entry Into the POLO Trial. J Clin Oncol. 2020 May 1;38(13):1442-1454. doi: 10.1200/JCO.19.01890. Epub 2020 Feb 19. PMID 32073954
- [Derived] Hammel P, Kindler HL, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Joo S, Yoo HK, Patel N, Golan T; POLO Investigators. Health-related quality of life in patients with a germline BRCA mutation and metastatic pancreatic cancer receiving maintenance olaparib. Ann Oncol. 2019 Dec 1;30(12):1959-1968. doi: 10.1093/annonc/mdz406. PMID 31562758
- [Derived] Lowery MA, Kelsen DP, Capanu M, Smith SC, Lee JW, Stadler ZK, Moore MJ, Kindler HL, Golan T, Segal A, Maynard H, Hollywood E, Moynahan M, Salo-Mullen EE, Do RKG, Chen AP, Yu KH, Tang LH, O'Reilly EM. Phase II trial of veliparib in patients with previously treated BRCA-mutated pancreas ductal adenocarcinoma. Eur J Cancer. 2018 Jan;89:19-26. doi: 10.1016/j.ejca.2017.11.004. Epub 2017 Dec 8. PMID 29223478
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081FC00001&attachmentIdentifier=9095e288-3d26-4c56-87dd-5dedc61f25c2&fileName=POLO_Revised_CSP_2-24Jul2019_Redacted.pdf&versionIdentifier=
- See also: Redacted_SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081FC00001&attachmentIdentifier=42f897a4-b682-4a0f-b2b0-cecf3f143423&fileName=D081FC00001_Redacted_SAP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081FC00001&attachmentIdentifier=adf11419-4145-42dc-bd0c-e36699d77c73&fileName=D081FC00001_CSR_SynopsisRedacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomised patients at a total of 59 study centres in 12 countries: United States of America (13), Germany (8), France (7), Israel (7), Spain (7), United Kingdom (6), Italy (4), Belgium (2), Republic of Korea (2), Australia (1), Canada (1) and Netherlands (1).
Pre-assignment Details: Screening Part 1 was only required if a patient's gBRCAm status was unknown and Screening Part 2 was for patients with known local germline BRCA (gBRCA) test. All other screening parameters were done as per the Study Schedule.
Groups:
- Olaparib 300 mg Twice Daily (bd): Randomised participants received orally 300 mg bd which were made up of 2 x 150 mg tablets bd with 100 mg tablets used to manage dose reductions.
- Placebo: Randomised participants received placebo tablets orally 300 mg bd which were made up of 2 x 150 mg tablets bd with 100 mg tablets used to manage dose reductions.
Period: Overall Study
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Started | 92 | 62
Completed | 19 | 7
Not Completed | 73 | 55
Not completed — Patient decision | 5 | 2
Not completed — Eligibility criteria not fulfilled | 0 | 1
Not completed — Death | 67 | 44
Not completed — Lost to Follow-up | 1 | 5
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set consisted of all randomised patients analysed on an intent to treat basis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo | Total
Number analyzed (Participants) | 92 | 62 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (10.27) | 56.4 (9.07) | 57.5 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 31 | 70
  Male | 53 | 31 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 88 | 60 | 148
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 82 | 59 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) by Blinded Independent Central Review (BICR) Using Modified Response Evaluation Criteria in Solid Tumours. This Study Used Modified RECIST Version (v) 1.1 (RECIST v1.1)
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo by PFS. The PFS was defined as the time from randomisation until the date of objective radiological disease progression according to modified RECIST v1.1 or death (by any cause in the absence of disease progression) regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to disease progression.
Time Frame: Up to 4 years
Population: Intention to treat (ITT): All randomised patients, Myriad confirmed Breast cancer susceptibility gene mutation (gBRCAm) subgroup.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 92 | 62
Months | 7.4 [4.14 to 11.01] | 3.8 [3.52 to 4.86]
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Superiority; p = 0.0038, Log-rank test; Hazard Ratio (HR) = 0.531, 95% CI 2-sided [0.346 to 0.815]

2. Secondary Outcome: Overall Survival (OS)
Description: To determine the efficacy by assessment of OS of olaparib maintenance monotherapy compared to placebo. The OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: Upto 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 92 | 62
Months | 19.0 [15.28 to 26.32] | 19.2 [14.32 to 26.12]
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Other; p = 0.3487, Log-rank test; Hazard Ratio (HR) = 0.831, 95% CI 2-sided [0.564 to 1.224]

3. Secondary Outcome: Time From Randomisation to Second Progression (PFS2)
Description: To determine efficacy by assessment of PFS2 of olaparib maintenance monotherapy compared to placebo. The PFS2 was defined as the time from the date of randomisation to the earliest of the progression event subsequent to that used for the primary variable PFS or death.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 92 | 62
Months | 16.9 [8.21 to 23.85] | 9.3 [8.15 to 13.54]
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Superiority; p = 0.0613, Log-rank test; Hazard Ratio (HR) = 0.659, 95% CI 2-sided [0.426 to 1.020]

4. Secondary Outcome: Time From Randomisation to Second Subsequent Therapy or Death (TSST)
Description: To determine the efficacy by assessment of TSST of olaparib maintenance monotherapy compared to placebo. The TSST was defined as time to second subsequent therapy or death.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 92 | 62
Months | 14.9 [9.13 to 19.78] | 9.6 [8.34 to 12.98]
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Superiority; p = 0.0111, Log-rank test; Hazard Ratio (HR) = 0.611, 95% CI 2-sided [0.418 to 0.894]

5. Secondary Outcome: Time From Randomisation to First Subsequent Therapy or Death (TFST)
Description: To determine the efficacy by assessment of TFST of olaparib maintenance monotherapy compared to placebo. The TFST was defined as time to first subsequent therapy or death.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 92 | 62
Months | 9.0 [6.21 to 12.85] | 5.4 [3.94 to 6.21]
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Superiority; p < 0.0001, Log-rank test; Hazard Ratio (HR) = 0.442, 95% CI 2-sided [0.297 to 0.658]

6. Secondary Outcome: Time From Randomisation to Study Treatment Discontinuation or Death (TDT)
Description: To determine the efficacy by assessment of TDT compared to placebo. compared to placebo. The TDT was defined as time to study treatment discontinuation or death.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 92 | 62
Months | 7.5 [5.52 to 10.97] | 3.8 [3.61 to 4.80]
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Superiority; p < 0.0001, Log-rank test; Hazard Ratio (HR) = 0.425, 95% CI 2-sided [0.289 to 0.627]

7. Secondary Outcome: Number of Participants With Objective Response Rate (ORR) by BICR Using Modified RECIST 1.1
Description: To determine efficacy by assessment of objective response rate according to modified RECIST 1.1 of olaparib maintenance monotherapy compared to placebo. The ORR is defined as the number of with a BoR of CR and PR according to the BICR data divided by the number of patients in the treatment group with measurable disease at baseline.
Time Frame: Up to 4 years
Population: All randomised patients with measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 72 | 49
Participants | 22 | 11
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Superiority; p = 0.3273, Regression, Logistic; Odds Ratio (OR) = 1.520, 95% CI 2-sided [0.668 to 3.610]

8. Secondary Outcome: Disease Control Rate (DCR) by BICR Using Modified RECIST 1.1
Description: Efficacy by assessment of disease control rate according to modified RECIST 1.1 of olaparib maintenance monotherapy compared to placebo.
Time Frame: At 16 weeks
Population: Intention to treat (ITT): All randomised patients
Measure: Number; unit: Participants
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 92 | 62
Participants
  Yes | 51 | 24
  No | 34 | 34
  Not evaluable/missing | 7 | 4

9. Secondary Outcome: Adjusted Mean Change From Baseline up to 6 Months in Global Quality of Life (QoL) Score From the EORTC-QLQ-C30 Questionnaire
Description: To assess the effect of olaparib on health-related quality of life (QoL) as measured by the EORTC-QLQ-C30 global QoL scale. The EORTC-QLQ-C30 is defined as EORTC QLQ-C30: a questionnaire (30 questions) used to evaluate disease symptoms, functional impacts (eg, physical functioning), and HRQoL and to characterize clinical benefit from the patient perspective. The HRQoL score ranges from 0 to 100.
  A higher score indicates better QoL. A score change of 10 points was pre-defined as clinically meaningful.
  bd twice daily.
Time Frame: From baseline up to 6 months
Population: Patient reported outcome (PRO) analysis set was defined as the analysis population for PRO data were a subset of the FAS (ITT) population who had evaluable baseline EORTC QLQ-C30 or QLQ-PAN26 forms where evaluable meant that at least 1 sub-scale baseline score could be determined from at least 1 of the 2 forms.
Measure: Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 84 | 55
Unit on scale | -1.03 [-3.826 to 1.759] | 1.18 [-2.585 to 4.939]
Statistical Analysis 1: Comparison: Olaparib 300 mg Twice Daily (bd) vs Placebo; Test type: Superiority; p = 0.355, Mixed Models Analysis; Mean Difference (Final Values) = -2.21, 95% CI 2-sided [-6.917 to 2.496]

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: To assess the safety and tolerability of olaparib maintenance monotherapy. SAE: serious adverse events CTCAE: Common Terminology Criteria for Adverse Events
Time Frame: Up to 4 years
Population: Safety Analysis Set consisted of all patients who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
Number analyzed (Participants) | 90 | 61
Participants
  Any AE | 89 | 56
  Any AE of CTCAE Grade 3 or higher | 44 | 15
  Any AE with outcome = death | 1 | 0
  Any SAE (including events with outcome = death) | 28 | 10
  AnyAE leading to withdrawal of olaparib/placebo | 8 | 1
  Any AE leading to dose interruption | 38 | 4
  Any AE leading to dose reduction | 16 | 3

ADVERSE EVENTS:
Time Frame: From informed consent until 30 days after last dose + subsequent treatment-related events reported (maximum up to 4 years).
Description: Only 90 patients in Olaparib and 61 patients in Placebo group were reported for safety because 3 patients did not receive study treatment and were not reported in the safety table.
Arm/Group | Olaparib 300 mg Twice Daily (bd) | Placebo
All-Cause Mortality (participants affected / at risk) | 68/92 | 52/62
Serious Adverse Events (participants affected / at risk) | 28/90 | 10/61
Other Adverse Events (participants affected / at risk) | 89/90 | 56/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib 300 mg Twice Daily (bd) (N=90) | Placebo (N=61)
Abdominal infection (Infections and infestations) | 1 | 0
Bartholinitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Vascular stenosis (Vascular disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Device occlusion (Product Issues) | 1 | 0
Stent malfunction (Product Issues) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Bronchiolitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olaparib 300 mg Twice Daily (bd) (N=90) | Placebo (N=61)
Nausea (Gastrointestinal disorders) | 44 (66) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 34 (49) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 26 (39) | 15 (17)
Constipation (Gastrointestinal disorders) | 25 (33) | 7 (8)
Vomiting (Gastrointestinal disorders) | 23 (49) | 9 (12)
Stomatitis (Gastrointestinal disorders) | 8 (10) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 9 (11) | 9 (10)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 9 (16) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 5 (6) | 6 (6)
Flatulence (Gastrointestinal disorders) | 2 (3) | 4 (4)
Fatigue (General disorders) | 42 (47) | 16 (19)
Asthenia (General disorders) | 16 (24) | 6 (6)
Pyrexia (General disorders) | 17 (28) | 4 (5)
Oedema peripheral (General disorders) | 8 (11) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (28) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (25) | 11 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (9) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Dysgeusia (Nervous system disorders) | 6 (6) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 9 (10) | 7 (7)
Dizziness (Nervous system disorders) | 8 (8) | 3 (4)
Headache (Nervous system disorders) | 8 (10) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 26 (35) | 10 (12)
Neutropenia (Blood and lymphatic system disorders) | 8 (9) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (9) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 24 (29) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (15) | 1/60 (1)
Rash (Skin and subcutaneous tissue disorders) | 12 (15) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11) | 4 (4)
Alanine aminotransferase increased (Investigations) | 10 (16) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (14) | 1 (1)
Blood creatinine increased (Investigations) | 7 (12) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 6 (7) | 3 (3)
Platelet count decreased (Investigations) | 5 (9) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 1 (1)
Anxiety (Psychiatric disorders) | 9 (10) | 2 (2)
Depression (Psychiatric disorders) | 5 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 2 (3)
Nasopharyngitis (Infections and infestations) | 12 (21) | 2 (2)
Influenza (Infections and infestations) | 6 (8) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 2 (2)
Influenza like illness (General disorders) | 6 (6) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 5 (9) | 0 (0)
Weight decreased (Investigations) | 7 (7) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 6 (9) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (16) | 0 (0)
Hypertension (Vascular disorders) | 5 (12) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This submission /document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT02184195/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT02184195/SAP_003.pdf